CLINICAL TRIAL: NCT02933697
Title: A Safety Study Assessing Oral Anticoagulation With Apixaban Versus Vitamin-K Antagonists in Patients With Atrial Fibrillation (AF) and End-Stage Kidney Disease (ESKD) on Chronic Hemodialysis Treatment
Brief Title: Compare Apixaban and Vitamin-K Antagonists in Patients With Atrial Fibrillation (AF) and End-Stage Kidney Disease (ESKD)
Acronym: AXADIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Atrial Fibrillation Network (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AXADIA - AFNET 8
Record Dates: First submitted 2016-10-07; First posted 2016-10-14 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation; End-stage Kidney Disease
Keywords: Atrial Fibrillation; Kidney disease; Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation; Kidney Failure, Chronic; Kidney Diseases | interventions — apixaban; Phenprocoumon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Active Comparator): 2.5 mg apixaban twice daily for 1 to 60 months
  Interventions: Drug: Apixaban
- Vitamin-K antagonists (Phenprocoumon) (Active Comparator): Phenprocoumon by INR (Target: 2.0-3.0) treatment for 1 to 60 months
  Interventions: Drug: Phenprocoumon

INTERVENTIONS:
Drug: Apixaban — Patients will be instructed to take one tablet of 2.5 mg twice daily: one tablet in the morning and one in the evening at approximately the same time every day (with about 12 hours gap) irrespective of the time of dialysis.
  Other Names: Eliquis
  Arms: Apixaban
Drug: Phenprocoumon — Subjects in phenprocoumon treatment group will receive phenprocoumon individually adjusted to an INR of 2.0-3.0 as recommended in the appropriate SmPC for AF patients.
  Other Names: Marcumar
  Arms: Vitamin-K antagonists (Phenprocoumon)

SUMMARY:
The Study is an open-labeled, randomized controlled trial, phase IIIb. Its objective is to assess the safety of the factor Xa inhibitor apixaban versus the vitamin-K antagonist (VKA) phenprocoumon in patients with NVAF and ESKD on hemodialysis. The safety will be assessed by means of the incidence of major and clinically relevant, non-major bleeding on anticoagulation.

DETAILED DESCRIPTION:
AXADIA is an investigator-driven, prospective, parallel-group, single country, multi-center phase IIIb trial to assess the safety of apixaban versus the vitamin-K antagonist phenprocoumon in patients with NVAF and ESKD on hemodialysis treatment. The trial will be conducted in about 25-30 sites in Germany.

The primary goal of this study is to assess the safety of two types of oral anticoagulants in patients with ESKD on hemodialysis with non-valvular atrial fibrillation (NVAF). The novel FXa inhibitor apixaban (at a reduced dose of 2x 2.5 mg/day) will be compared to the vitamin-K antagonist (VKA) phenprocoumon (target range: International Normalized Ratio (INR) 2.0-3.0) regarding bleeding rates during chronic administration for prevention of stroke or systemic embolism.

The primary hypothesis of the study is that oral anticoagulation with apixaban will improve the safety by significantly reducing bleeding rates in patients with ESKD on hemodialysis and NVAF compared to the VKA phenprocoumon.

ELIGIBILITY:
Inclusion Criteria:

* End-stage kidney disease (ESKD) with chronic hemodialysis treatment 3 times per week (with about at least 3.5 hours per dialysis)
* Chronic (i.e. repeated) paroxysmal, persistent or permanent atrial fibrillation (AF) or atrial flutter (AFL) documented by standard or Holter ECG on at least 2 separate days before (or apart from) hemodialysis procedures
* Increased risk of stroke or systemic embolism identified by a CHA2DS2-VASc score of 2 or more as an indication for oral anticoagulation
* Patients with ischemic stroke that meet the above criteria, can be included after more than 3 months if not severely handicapped (modified Rankin scale 0 or 1 of 6, i.e. no symptoms or no significant disability and able to carry out all usual activities, despite some symptoms (Farrell, Godwin, Richards, and Warlow (1991))
* Males and females, aged 18 or older

Exclusion Criteria:

* AF or AFL due to reversible causes (e.g., thyrotoxicosis, pericarditis)
* Patients with a new onset of hemodialysis within the last 3 months
* Clinically significant (moderate or severe) aortic and mitral stenosis
* Conditions other than AF or AFL that require chronic anticoagulation (e.g., a prosthetic mechanical heart valve).
* Active infective endocarditis
* Any planned interventional or surgical AF or AFL ablation procedure
* Any active bleeding
* A serious bleeding event in the previous 6 months before screening
* Inadequately controlled (HbA1c levels >8.5%) or untreated diabetes
* History of malignant neoplasms at high risk of current bleeding (see summary of product characteristics (SmPC) of study drugs)
* Known indication for treatment with NSAIDs (see SmPC of study drugs) - acetylsalicylic acid (ASA) up to 100 mg per day is allowed
* Known Antiphospholipid Syndrome requiring anticoagulation
* Impaired liver function e.g., caused by active infection with HIV, HBV or HCV, hepatitis or other liver damage (No limits for ALT and AST values are defined in this study protocol, although mentioned in the SmPC because they are frequently elevated in dialysis patients. In case of clinically relevant increase of ALT or AST level, patient's eligibility is to be decided by the responsible investigator)
* Any type of stroke within 3 months prior to baseline
* Other indication for anticoagulation than AF or AFL
* Valvular heart disease requiring surgery
* A high risk of bleeding (e.g., active peptic ulcer disease, a platelet count of <100,000 per cubic millimeter or hemoglobin level of <8 g per deciliter)
* Documented hemorrhagic tendencies or blood dyscrasias
* Current alcohol or drug abuse
* Life expectancy of less than 1 year
* Indication for dual platelet inhibition at baseline (ASA ≤ 100 mg/day is allowed, clopidrogel is excluded at any dose).
* Active infection or symptoms suggestive of COVID-19 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Assess the safety of the factor Xa inhibitor apixaban versus a vitamin-K antagonist phenprocoumon in patients with NVAF and ESKD on hemodialysis. | 1-60 months
  The safety will be assessed by means of the incidence of major and clinically relevant, non-major bleeding as well as specific bleedings in dialysis patients (e.g., after shunt removal) on anticoagulation.

SECONDARY OUTCOMES:
Compare the efficacy of the factor Xa inhibitor apixaban with the VKA phenprocoumon regarding prevention of thromboembolic events in patients with ESKD on hemodialysis and AF | 1-60 months
  The efficacy of the factor Xa inhibitor apixaban with the VKA phenprocoumon regarding prevention of thromboembolic events in patients with ESKD on hemodialysis and AF

CONTACTS AND LOCATIONS:
Overall Officials: Holger Reinecke, Prof. Dr., Principal Investigator — Universitätsklinikum Münster
Locations (1):
- Universitätsklinikum Münster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinecke H, Engelbertz C, Bauersachs R, Breithardt G, Echterhoff HH, Gerss J, Haeusler KG, Hewing B, Hoyer J, Juergensmeyer S, Klingenheben T, Knapp G, Christian Rump L, Schmidt-Guertler H, Wanner C, Kirchhof P, Goerlich D. A Randomized Controlled Trial Comparing Apixaban With the Vitamin K Antagonist Phenprocoumon in Patients on Chronic Hemodialysis: The AXADIA-AFNET 8 Study. Circulation. 2023 Jan 24;147(4):296-309. doi: 10.1161/CIRCULATIONAHA.122.062779. Epub 2022 Nov 6. PMID 36335915
- [Derived] Reinecke H, Jurgensmeyer S, Engelbertz C, Gerss J, Kirchhof P, Breithardt G, Bauersachs R, Wanner C. Design and rationale of a randomised controlled trial comparing apixaban to phenprocoumon in patients with atrial fibrillation on chronic haemodialysis: the AXADIA-AFNET 8 study. BMJ Open. 2018 Sep 10;8(9):e022690. doi: 10.1136/bmjopen-2018-022690. PMID 30206088